CLINICAL TRIAL: NCT05729256
Title: Alcohol and "Heat of the Moment" Sexual Decision Making Among MSM: Identifying Mechanisms of Sexual Risk and Promoting Behavior Change Through Brief Intervention
Brief Title: Alcohol and "Heat of the Moment" Sexual Decision Making
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: Syracuse University (Other); University of South Dakota (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 6603e; R01AA030461-01 (NIH)
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Alcohol Drinking; Sex, Unsafe; Hiv
MeSH Terms: conditions — Alcohol Drinking; Unsafe Sex; Acquired Immunodeficiency Syndrome | interventions — Crisis Intervention

STUDY DESIGN:
Intervention Model Description: Participants randomly assigned to either intervention or control
Who Masked: Outcomes Assessor
Masking Description: Trial procedures designed so that the post-intervention assessor is blind to condition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Regulation Intervention (Experimental): Single session motivational intervention on reducing heavy drinking and sexual risk behavior, encouraging consideration of pre-exposure prophylaxis (PrEP), followed by 4 weeks of text messages on content relevant to drinking goals and support for healthy sexual choices
  Interventions: Behavioral: Self-Regulation Intervention
- Brief Advice and Information (Active Comparator): Single session to provide psychoeducation about heavy drinking risks, discussion of barriers to safe sex, information about pre-exposure prophylaxis (PrEP)
  Interventions: Behavioral: Brief Advice and Information

INTERVENTIONS:
Behavioral: Self-Regulation Intervention — Single session motivational intervention on reducing heavy drinking and sexual risk behavior, encouraging consideration of pre-exposure prophylaxis (PrEP), followed by 4 weeks of text messages on content relevant to drinking goals and support for healthy sexual choices
  Arms: Self-Regulation Intervention
Behavioral: Brief Advice and Information — Psychoeducation about heavy drinking risks, discussion of barriers to safe sex, information about pre-exposure prophylaxis (PrEP)
  Arms: Brief Advice and Information

SUMMARY:
HIV transmission remains a significant public health concern, especially among men who have sex with men (MSM). Condomless anal intercourse (CAI) continues to be the major route of transmission for MSM. Thus, to reduce the incidence of HIV, it is critical to identify how contextual risk factors influence CAI and develop behavioral strategies that modify risk factors directly or reduce their influence on behavior. This study will examine the mechanisms through which one of the central contextual risk factors, heavy drinking, influences sexual decision processes in the natural environment and test the benefit of a brief intervention designed to reduce sexual risk behavior among those who engage in heavy drinking.

DETAILED DESCRIPTION:
Despite prevention efforts over the past two decades, HIV transmission remains a significant public health concern, especially among men who have sex with men (MSM). Approximately 65% of new HIV diagnoses in the United States are due to male-to-male sexual contact. Condomless anal intercourse (CAI) continues to be the major route of transmission for MSM. Thus, to reduce the incidence of HIV, it is critical to identify risk factors that underlie HIV acquisition and transmission and develop behavioral strategies that modify them directly or reduce the influence of these factors on behavior. Alcohol use, particularly heavy episodic drinking, is a central modifiable risk factor that may increase CAI in conjunction with other contextual variables. Although there have been a limited number of HIV prevention interventions that incorporate alcohol in sexual risk reduction efforts, relatively little is known about how such interventions impact sexual decision-making in "heat-of the-moment", particularly while intoxicated and in high arousal states that commonly are proximal to sexual behavior.

The goals of this study are to: (1) better understand the within-person mechanisms linking alcohol and arousal with CAI and (2) test the efficacy of an HIV prevention intervention approach that both reduces alcohol consumption and mitigate the influence of intoxication and arousal on CAI. These complementary objectives are addressed through an experience sampling method study (ESM) that examines the impact of an HIV prevention intervention that targets sexual risk and alcohol use. This study will examine whether mechanisms that underlie sexual risk in the natural environment and can be modified by intervention.

In the proposed study, non-monogamous adult MSM who engage in heavy drinking and CAI will be randomly assigned to an intervention condition that addresses alcohol use and sexual decision-making in "heat-of-the-moment" situations. The intervention will be preceded and followed by 3-week ESM bursts of intensive longitudinal assessment of alcohol use, arousal, sexual delay discounting, working memory, and CAI. 4-month follow-up data will be collected. Results will contribute to the long-term goal of enhancing effectiveness of behavioral HIV prevention interventions that address alcohol use.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Cisgender man who has had condomless anal intercourse with another man in the past 3 months
* Engaged in heavy drinking (assessed by either weekly National Institute on Alcohol Abuse and Alcoholism guidelines [> 14 for men], and/or a heavy drinking episode in the past month [> 4 drinks on an occasion])
* Has a smartphone

Exclusion Criteria:

* HIV-infection
* Currently using PrEP
* In an exclusive monogamous sexual relationship
* History of bipolar disorder, schizophrenia, other psychotic disorder, or current suicidal intent
* Current treatment for alcohol use disorder or substance use disorder
* Unable to provide one or more individuals who can serve as an alternate contact

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender men
Enrollment: 354 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Count of number of times engaged in Condomless Anal Intercourse (CAI) from Sexual Behavior Survey | Past 90 days
  Self-reported number of times engaged in CAI
Heavy Drinking Episodes from the Quick Drinking Screen | Past 90 days
  Self-reported number of days consumed 5 or more standard drinks
Average number of drinks per week from the Quick Drinking Screen | Past 90 days
  Self-reported average number of drinks per week multiplied by frequency of drinking per week
Condomless Anal Intercourse: Experience Sampling | ESM assessments over a 3 week period
  Self-reported frequency of CAI from experience sampling questions
Alcohol Use: Experience Sampling | ESM assessments over 3 week period
  Self-reported number of drinks and perceived intoxication (composite variable)

CONTACTS AND LOCATIONS:
Overall Officials: Tibor Palfai, PhD, Principal Investigator — Boston University
Locations (1):
- Boston University Department of Psychological and Brain Sciences, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared following release within one year of the trial end to investigators who make specific requests in writing regarding analysis plans. Plans will be reviewed with co-investigators to ensure that there is no overlap with planned analyses. Specific de-identified data set will be provided to other researchers after this review.
  In addition, data will be shared according to the guidelines for the National Institute of Mental Health Data Archive (NDA)
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available one year after the end of the study. Support will be provided for data access for up to 5 years.
Access Criteria: Based on review of data plan from the Multiple Principal Investigators of the study

REFERENCES:
- [Background] Sobell LC, Agrawal S, Sobell MB, Leo GI, Young LJ, Cunningham JA, Simco ER. Comparison of a quick drinking screen with the timeline followback for individuals with alcohol problems. J Stud Alcohol. 2003 Nov;64(6):858-61. doi: 10.15288/jsa.2003.64.858. PMID 14743950
- [Background] Gordon CM, Carey MP, Carey KB. Effects of a drinking event on behavioral skills and condom attitudes in men: implications for HIV risk from a controlled experiment. Health Psychol. 1997 Sep;16(5):490-5. doi: 10.1037//0278-6133.16.5.490. PMID 9302547